CLINICAL TRIAL: NCT05168657
Title: Assessing Feasibility, Safety, and Efficacy of Deploying a Closed-loop Automated Insulin Delivery System by Community-based Primary Care Physicians and Academic Endocrinologists, in Person and Through Telehealth
Brief Title: Feasibility of Closed-loop Automated Insulin Delivery System by Primary Care & Endocrinology, in Person & Via Telehealth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Beta Bionics, Inc. (Industry); Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 21-3272
Record Dates: First submitted 2021-11-23; First posted 2021-12-23 (Actual); Results first posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Diabetes Mellitus, Type 1; Type 1 Diabetes; Diabetes, Autoimmune; Diabetes type1; Autoimmune Diabetes; Diabetes Mellitus, Brittle; Diabetes Mellitus, Insulin-Dependent; Diabetes Mellitus, Insulin-Dependent, 1; Diabetes Mellitus, Juvenile-Onset; Diabetes Mellitus, Ketosis-Prone; Diabetes Mellitus, Sudden-Onset; Insulin-Dependent Diabetes Mellitus 1; Juvenile-Onset Diabetes; Type 1 Diabetes Mellitus
Keywords: bionic pancreas; closed loop; insulin; Pancreas, Artificial; automated insulin delivery system; t1d; t1dm
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Random-order cross over trial in a home-use setting with two 14-day study arms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (8):
- EN-IP-UC first, Then BP (Experimental): Random-order cross-over participants managed by ENDOCRINOLOGY with IN-PERSON visits, assigned by randomization to undergo 14 days of Usual Care, followed by 14 days of Bionic Pancreas. There was no washout period between arms.
  Interventions: Other: Usual Care
- EN-TH-UC first, Then BP (Experimental): Random-order cross-over participants managed by ENDOCRINOLOGY with TELEHEALTH visits, assigned by randomization to undergo 14 days of Usual Care, followed by 14 days of Bionic Pancreas. There was no washout period between arms.
  Interventions: Other: Usual Care
- EN-IP-BP first, Then UC (Experimental): Random-order cross-over participants managed by ENDOCRINOLOGY with IN PERSON visits, assigned by randomization to undergo 14 days of Bionic Pancreas, followed by 14 days of Usual Care. There was no washout period between arms.
  Interventions: Device: Bionic Pancreas
- EN-TH-BP first, Then UC (Experimental): Random-order cross-over participants managed by ENDOCRINOLOGY with TELEHEALTH visits, assigned by randomization to undergo 14 days of Bionic Pancreas, followed by 14 days of Usual Care. There was no washout period between arms.
  Interventions: Device: Bionic Pancreas
- PC-IP-UC first, Then BP (Experimental): Random-order cross-over participants managed by PRIMARY CARE with IN-PERSON visits, assigned by randomization to undergo 14 days of Usual Care, followed by 14 days of Bionic Pancreas. There was no washout period between arms.
  Interventions: Other: Usual Care
- PC-TH-UC first, Then BP (Experimental): Random-order cross-over participants managed by PRIMARY CARE with TELEHEALTH visits, assigned by randomization to undergo 14 days of Usual Care, followed by 14 days of Bionic Pancreas. There was no washout period between arms.
  Interventions: Other: Usual Care
- PC-IP-BP first, Then UC (Experimental): Random-order cross-over participants managed by PRIMARY CARE with IN PERSON visits, assigned by randomization to undergo 14 days of Bionic Pancreas, followed by 14 days of Usual Care. There was no washout period between arms.
  Interventions: Device: Bionic Pancreas
- PC-TH-BP first, Then UC (Experimental): Random-order cross-over participants managed by PRIMARY CARE with TELEHEALTH visits, assigned by randomization to undergo 14 days of Bionic Pancreas, followed by 14 days of Usual Care. There was no washout period between arms.
  Interventions: Device: Bionic Pancreas

INTERVENTIONS:
Device: Bionic Pancreas — 14 days using the insulin-only configuration of the iLet Bionic Pancreas (Beta Bionics, Inc.), which automates insulin delivery, as the only intended mode of insulin delivery.
  Other Names: BP
  Arms: EN-IP-BP first, Then UC; EN-TH-BP first, Then UC; PC-IP-BP first, Then UC; PC-TH-BP first, Then UC
Other: Usual Care — 14 days of the participant's usual care of their type 1 diabetes
  Other Names: UC
  Arms: EN-IP-UC first, Then BP; EN-TH-UC first, Then BP; PC-IP-UC first, Then BP; PC-TH-UC first, Then BP

SUMMARY:
This is a study assessing the feasibility of using the insulin-only configuration of the iLet bionic pancreas with initiation in pump-naïve people with type 1 diabetes in a primary care practice with either in-person training and follow-up (PC-IP) or with training and follow-up via telehealth (PC-TH). As a comparison, the iLet will be initiated by an academic endocrinology practice with either in-person training and follow-up (EN-IP) or with training and follow-up via telehealth (EN-TH).

DETAILED DESCRIPTION:
This is a study assessing the feasibility of deploying the iLet bionic pancreas system in the insulin-only configuration to pump-naïve MDI users with type 1 diabetes, in the setting of being recruited from community-based primary care practices and being trained and managed by primary care providers (PC group), and in pump- and CGM-experienced (sensor-augmented pump or hybrid closed-loop) users with type 1 diabetes recruited from, trained, and managed by an academic endocrinology practice (EN group). In both practice settings, the exclusive use of telehealth (TH) visits will be assessed, as will the use of in-person (IP) visits. We will enroll 40 adult volunteers (≥ 18 years old) with type 1 diabetes, 20 who are insulin pump naïve MDI users enrolled from community primary care practices by University of Colorado Family Medicine (PC group) and 20 who are technology-savvy sensor-augmented pump or hybrid closed-loop users enrolled by the Massachusetts General Hospital Diabetes Clinical Research Center (EN group). Ten of the participants at each center will be trained and managed throughout the trial using in-person visits (PC-IP and EN-IP groups) and the other ten from each center will be trained and managed throughout the trial exclusively via telehealth visits (PC-TH and EN-TH groups). This will result in four study cohorts overall (endocrinology in-person, endocrinology telehealth, primary care in-person, primary care telehealth). Subjects in all four groups will each participate, in random order, in one 14-day study arm under their own usual care (UC arm) and one 14-day study arm under the insulin-only configuration of the iLet bionic pancreas (iLet arm).

ELIGIBILITY:
Inclusion Criteria

1. Age 18-85 years, BMI ≥ 18.5, have had clinical type 1 diabetes for at least one year, and have taken insulin for at least 1 year

   1. Prescription diabetes medication regimen stable for > 1 month, including any adjunctive anti-diabetic medications (except for medications that will not affect the safety of the study and are not expected to affect any outcome of the study, in the judgment of the site principal investigator)
   2. This does not include changes to any insulin doses, including basal rates/long-acting insulin doses, carbohydrate to insulin ratios and correction factors
2. Willing to wear one Dexcom CGM transmitter and sensor (sensor must be changed every 10 days), and one infusion set that must be replaced at least every 3 days.
3. Endocrinology practice criterion is that diabetes is managed using sensor-augmented insulin pump therapy or artificial pancreas therapy for ≥ 3 months)
4. Primary care practice criteria are that diabetes is managed by multiple daily insulin injections (insulin-pump naïve).
5. TH group criterion is that participant must have hardware and internet access capable of 2-way video and audio communication

Exclusion Criteria

1. Unable to provide informed consent (e.g. impaired cognition or judgment)
2. Unable to safely comply with study procedures and reporting requirements (e.g. impairment of vision or dexterity that prevents safe operation of the bionic pancreas, impaired memory)
3. Unable to speak and read English, as iLet BP support materials and device menus are currently available in English only.
4. Plan to change usual diabetes regimen in the next 3 months including before and during participation in the study

   1. This would include changing from MDI to pump or from pump to MDI, and starting a CGM if not previously used
   2. This would not include changes to any insulin doses, including basal rates/long acting insulin doses, carbohydrate to insulin ratios and correction factors
5. Current use of non-FDA approved closed-loop or hybrid closed-loop insulin delivery system (e.g. "Loop" or "Open APS")
6. Unwilling to switch to lispro or aspart for the duration of the study's iLet arm (e.g. from Fiasp or Lyumjev)
7. Known hemoglobinopathy (sickle cell trait is not an exclusion)
8. Current participation in another diabetes-related clinical trial, has a medical condition, or use of a medication that, in the judgment of the investigator, could compromise the results of this study or the safety of the participant
9. History of diabetes due to cystic fibrosis, pancreatitis, or other pancreatic disease, including pancreatic tumor or insulinoma, or history of complete pancreatectomy
10. Have a history of intermittently required glucocorticoid treatment (e.g., but not limited to, for the treatment of asthma, inflammatory bowel disease).
11. A1c >11.0% (most recent value up to 1 year prior acceptable; if none available or >1 year prior, participant will be instructed to obtain A1c through their usual care provider and to make copy of result available to study team)
12. History of diabetic ketoacidosis (DKA) within the past month
13. Electrically powered implants (e.g. cochlear implants, neurostimulators) that might be susceptible to RF interference
14. Established history of allergy or severe reaction to adhesive or tape that must be used in the study
15. Currently treated with GLP-1 analogue, thiazolidinedione (TZD), sulfonylurea, pramlintide, or SGLT-2 inhibitor medication (use more than 3 months prior to enrollment is acceptable)

    a. If using metformin, participants: i. Must be on a stable dose for 1 month prior to enrollment ii. Metformin can be continued while the iLet is used
16. Pregnant (positive urine HCG), breast feeding, plan to become pregnant in the next 6 months, or premenopausal participants who are sexually active without use of contraception
17. Renal failure on dialysis or chronic renal disease with a GFR or eGFR <30mL/min (values within the last two years will be accepted; if none available or >2 years prior, participant will be instructed to obtain GFR or eGFR through their usual care provider and to make copy of result available to study team)
18. Any condition that, in the opinion of the site principal investigator, could interfere with the safe or effective completion of the study.

    a. Conditions to be considered by the investigator may include, but are not limited to, the following: i. Alcohol or drug abuse ii. Use of prescription drugs that may dull the sensorium, reduce sensitivity to symptoms of hypoglycemia, or hinder decision making during the period of participation in the study iii. Coronary artery disease that is not stable with medical management, including unstable angina, angina that prevents moderate exercise (e.g. exercise of intensity up to 6 METS) despite medical management, or within the last 12 months before screening, a history of myocardial infarction, percutaneous coronary intervention, enzymatic lysis of a presumed coronary occlusion, or coronary artery bypass grafting iv. Known history of prolonged QTc interval, malignant arrhythmia, or congenital heart disease v. Congestive heart failure with New York Heart Association (NYHA) Functional Classification III or IV vi. History of TIA or stroke in the last 12 months vii. Untreated or inadequately treated mental illness viii. History of eating disorder within the last 2 years, such as anorexia, bulimia, or diabulimia or omission of insulin to manipulate weight ix. History of intentional, inappropriate administration of insulin leading to severe hypoglycemia requiring treatment
19. Employed by, or having immediate family members employed by Beta Bionics, or being directly involved in conducting the clinical trial, or having a direct supervisor at place of employment who is also directly involved in conducting the clinical trial (as a study investigator, coordinator, etc.); or having a first-degree relative who is directly involved in conducting the clinical trial
20. Unable to avoid hydroxyurea for duration of study (interferes with accuracy of Dexcom G6 CGM)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean M Oser, MD, MPH, Principal Investigator — University of Colorado, Denver; Tamara K Oser, MD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Deidentified glucose data and psychosocial data will be shared with research collaborators.
Supporting Information: Study Protocol

RESULTS

PARTICIPANT FLOW:
Groups:
- EN-IP-BP First, Then UC; PC-IP-BP First, Then UC: Random-order cross-over participants managed by ENDOCRINOLOGY with IN-PERSON visits, assigned by randomization to undergo 14 days of Bionic Pancreas, followed by 14 days of Usual Care. There was no washout period between arms.
  Usual Care: 14 days of the participant's usual care of their type 1 diabetes
- EN-TH-BP First, Then UC; PC-TH-BP First, Then BP: Random-order cross-over participants managed by ENDOCRINOLOGY with TELEHEALTH visits, assigned by randomization to undergo 14 days of Bionic Pancreas, followed by 14 days of Usual Care. There was no washout period between arms.
  Usual Care: 14 days of the participant's usual care of their type 1 diabetes
- PC-IP-UC First, Then BP: Random-order cross-over participants managed by ENDOCRINOLOGY with IN-PERSON visits, assigned by randomization to undergo 14 days of Usual Care, followed by 14 days of Bionic Pancreas. There was no washout period between arms.
  Usual Care: 14 days of the participant's usual care of their type 1 diabetes
- PC-TH-UC First, Then BP: Random-order cross-over participants managed by ENDOCRINOLOGY with TELEHEALTH visits, assigned by randomization to undergo 14 days of Usual Care, followed by 14 days of Bionic Pancreas. There was no washout period between arms.
  Usual Care: 14 days of the participant's usual care of their type 1 diabetes
Period: Overall Study
Arm/Group | EN-IP-UC First, Then BP | EN-TH-UC First, Then BP | EN-IP-BP First, Then UC | EN-TH-BP First, Then UC | PC-IP-UC First, Then BP | PC-TH-UC First, Then BP | PC-IP-BP First, Then UC | PC-TH-BP First, Then BP
Started | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 4 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- EN-IP: Random-order cross-over participants on BIONIC PANCREAS managed by ENDOCRINOLOGY with IN PERSON visits. Participants will be randomly assigned to initiate trial participation with either Bionic Pancreas intervention or Usual Care intervention, followed by the other intervention. Each intervention will consist of 14 days.
  Bionic Pancreas: 14 days using the insulin-only configuration of the iLet Bionic Pancreas (Beta Bionics, Inc.), which automates insulin delivery, as the only intended mode of insulin delivery.
- EN-TH: Random-order cross-over participants on BIONIC PANCREAS managed by ENDOCRINOLOGY with TELEHEALTH visits. Participants will be randomly assigned to initiate trial participation with either Bionic Pancreas intervention or Usual Care intervention, followed by the other intervention. Each intervention will consist of 14 days.
  Bionic Pancreas: 14 days using the insulin-only configuration of the iLet Bionic Pancreas (Beta Bionics, Inc.), which automates insulin delivery, as the only intended mode of insulin delivery.
  Telehealth: Study participation will be managed via telehealth visits.
- PC-IP: Random-order cross-over participants on BIONIC PANCREAS managed by PRIMARY CARE with IN PERSON visits. Participants will be randomly assigned to initiate trial participation with either Bionic Pancreas intervention or Usual Care intervention, followed by the other intervention. Each intervention will consist of 14 days.
  Bionic Pancreas: 14 days using the insulin-only configuration of the iLet Bionic Pancreas (Beta Bionics, Inc.), which automates insulin delivery, as the only intended mode of insulin delivery.
- PC-TH: Random-order cross-over participants on BIONIC PANCREAS managed by PRIMARY CARE with TELEHEALTH visits. Participants will be randomly assigned to initiate trial participation with either Bionic Pancreas intervention or Usual Care intervention, followed by the other intervention. Each intervention will consist of 14 days.
  Bionic Pancreas: 14 days using the insulin-only configuration of the iLet Bionic Pancreas (Beta Bionics, Inc.), which automates insulin delivery, as the only intended mode of insulin delivery.
  Telehealth: Study participation will be managed via telehealth visits.
- Total: Total of all reporting groups
Arm/Group | EN-IP | EN-TH | PC-IP | PC-TH | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 8 | 9 | 36
  >=65 years | 0 | 1 | 2 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (15.3) | 45.7 (12.3) | 44.6 (13.5) | 44.4 (16.7) | 44.8 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 4 | 3 | 17
  Male | 4 | 6 | 6 | 7 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 10 | 10 | 8 | 9 | 37
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 9 | 10 | 9 | 6 | 34
  More than one race | 0 | 0 | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 10 | 40
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.3 (5.3) | 29.4 (4.4) | 25.8 (2.8) | 27.5 (4.9) | 27.5 (4.5)
HbA1c [Mean (Standard Deviation); unit: % (of hemoglobin that is glycosylated] | 7.3 (1.1) | 7.2 (0.3) | 6.8 (0.6) | 7.0 (1.1) | 7.1 (0.8)
Diabetes duration [Mean (Standard Deviation); unit: years] | 26.4 (15.8) | 31.5 (10.9) | 15.2 (12.3) | 21.3 (16.0) | 23.6 (14.7)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Individuals With Mean CGM Glucose <183 mg/dL (Corresponding to an Estimated HbA1c of <8.0%) on Days 3-14, by Group.
Description: The outcome is categorical, and the primary outcome is not a direct comparison of the mean CGM glucose between the groups.
Time Frame: BP Arm Days 3-14
Population: Our primary outcome measure is restricted to the BP arm only, as pre-specified in the protocol. UC arm data is not relevant to this measure. One EN-IP participant was excluded from analysis because they withdrew from the study before beginning the BP arm; therefore 9 rather than 10 participants were included in the analysis for this group.
Measure: Number; unit: percentage of participants
Arm/Group | EN-IP | EN-TH | PC-IP | PC-TH
Number analyzed (Participants) | 9 | 10 | 10 | 10
percentage of participants | 89 | 100 | 100 | 100

2. Secondary Outcome: Mean CGM Glucose on Days 3-14
Description: Individual CGM values from days 3-14 were averaged together for each participant.
Time Frame: BP Arm Days 3-14
Population: This secondary outcome measure is restricted to the BP arm only, as pre-specified in the protocol. UC arm data is not relevant to this measure. One EN-IP participant was excluded from analysis because they withdrew from the study before beginning the BP arm; therefore 9 rather than 10 participants were included in the analysis for this group.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | EN-IP | EN-TH | PC-IP | PC-TH
Number analyzed (Participants) | 9 | 10 | 10 | 10
mg/dL | 155.9 (56.3) | 152.5 (52.2) | 145.0 (48.0) | 152.6 (44.8)

3. Secondary Outcome: Percentage of Time With CGM Glucose <54 mg/dl on Days 3-14
Description: Calculated from all individual CGM values from days 3-14 for each participant.
Time Frame: BP Arm Days 3-14
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percentage of time
Groups:
- EN-IP: Random-order cross-over participants on BIONIC PANCREAS managed by ENDOCRINOLOGY with IN PERSON visits. Participants will be randomly assigned to initiate trial participation with either Bionic Pancreas intervention or Usual Care intervention, followed by the other intervention. Each intervention will consist of 14 days.
- EN-TH: Random-order cross-over participants on BIONIC PANCREAS managed by ENDOCRINOLOGY with TELEHEALTH visits. Participants will be randomly assigned to initiate trial participation with either Bionic Pancreas intervention or Usual Care intervention, followed by the other intervention. Each intervention will consist of 14 days.
- PC-IP: Random-order cross-over participants on BIONIC PANCREAS managed by PRIMARY CARE with IN PERSON visits. Participants will be randomly assigned to initiate trial participation with either Bionic Pancreas intervention or Usual Care intervention, followed by the other intervention. Each intervention will consist of 14 days.
- PC-TH: Random-order cross-over participants on BIONIC PANCREAS managed by PRIMARY CARE with TELEHEALTH visits. Participants will be randomly assigned to initiate trial participation with either Bionic Pancreas intervention or Usual Care intervention, followed by the other intervention. Each intervention will consist of 14 days.
Arm/Group | EN-IP | EN-TH | PC-IP | PC-TH
Number analyzed (Participants) | 9 | 10 | 10 | 10
percentage of time | 0.48 [0.17 to 0.97] | 0.18 [0.00 to 0.95] | 0.14 [0.06 to 0.43] | 0.00 [0.00 to 0.30]

4. Secondary Outcome: Percentage of Time With CGM Glucose in the 70-180 mg/dl Range on Days 3-14
Description: Calculated from all individual CGM values from days 3-14 for each participant.
Time Frame: BP Arm Days 3-14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | EN-IP | EN-TH | PC-IP | PC-TH
Number analyzed (Participants) | 9 | 10 | 10 | 10
percentage of time | 67.9 (10.8) | 71.6 (5.0) | 78.6 (10.2) | 75.1 (8.6)

5. Secondary Outcome: Percentage of Individuals With Mean CGM Glucose <154 mg/dL (Corresponding to an Estimated HbA1c of <7.0%) on Days 3-14, by Group.
Description: Calculated from all individual CGM values from days 3-14 for each participant.
Time Frame: BP Arm Days 3-14
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | EN-IP | EN-TH | PC-IP | PC-TH
Number analyzed (Participants) | 9 | 10 | 10 | 10
percentage of participants | 67 | 50 | 80 | 60

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for each participant from the time of their enrollment through completion of the study, resolution of any adverse events if applicable, or until lost to follow-up. This ranged from approximately 30 days to 4 months, per participant.
Description: Adverse events were assessed systematically at each participant visit following enrollment and non-systematically via self-report. One EN-IP-BP participant withdrew from the study before beginning the BP arm; therefore 4 rather than 5 participants were at-risk for this group.
Groups:
- PC Pre-randomization: Random-order cross-over participants managed by PRIMARY CARE who were not yet randomized.
- EN Pre-randomization: Random-order cross-over participants managed by ENDOCRINOLOGY who were not yet randomized.
- PC-IP-UC: Random-order cross-over participants managed by PRIMARY CARE with IN-PERSON visits, assigned by randomization to undergo 14 days of Usual Care, followed by 14 days of Bionic Pancreas. There was no washout period between arms.
  Usual Care: 14 days of the participant's usual care of their type 1 diabetes.
- PC-IP-BP: Random-order cross-over participants managed by PRIMARY CARE with IN-PERSON visits, assigned by randomization to undergo 14 days of Bionic Pancreas, followed by 14 days of Usual Care. There was no washout period between arms.
  Bionic Pancreas: 14 days using the insulin-only configuration of the iLet Bionic Pancreas (Beta Bionics, Inc.), which automates insulin delivery, as the only intended mode of insulin delivery.
- PC-TH-UC: Random-order cross-over participants managed by PRIMARY CARE with TELEHEALTH visits, assigned by randomization to undergo 14 days of Usual Care, followed by 14 days of Bionic Pancreas. There was no washout period between arms.
  Usual Care: 14 days of the participant's usual care of their type 1 diabetes.
- PC-TH-BP: Random-order cross-over participants managed by PRIMARY CARE with TELEHEALTH visits, assigned by randomization to undergo 14 days of Bionic Pancreas, followed by 14 days of Usual Care. There was no washout period between arms.
  Bionic Pancreas: 14 days using the insulin-only configuration of the iLet Bionic Pancreas (Beta Bionics, Inc.), which automates insulin delivery, as the only intended mode of insulin delivery.
- EN-IP-UC: Random-order cross-over participants managed by ENDOCRINOLOGY with IN-PERSON visits, assigned by randomization to undergo 14 days of Usual Care, followed by 14 days of Bionic Pancreas. There was no washout period between arms.
  Usual Care: 14 days of the participant's usual care of their type 1 diabetes.
- EN-IP-BP: Random-order cross-over participants managed by ENDOCRINOLOGY with IN-PERSON visits, assigned by randomization to undergo 14 days of Bionic Pancreas, followed by 14 days of Usual Care. There was no washout period between arms.
  Bionic Pancreas: 14 days using the insulin-only configuration of the iLet Bionic Pancreas (Beta Bionics, Inc.), which automates insulin delivery, as the only intended mode of insulin delivery.
- EN-TH-UC: Random-order cross-over participants managed by ENDOCRINOLOGY with TELEHEALTH visits, assigned by randomization to undergo 14 days of Usual Care, followed by 14 days of Bionic Pancreas. There was no washout period between arms.
  Usual Care: 14 days of the participant's usual care of their type 1 diabetes.
- EN-TH-BP: Random-order cross-over participants managed by ENDOCRINOLOGY with TELEHEALTH visits, assigned by randomization to undergo 14 days of Bionic Pancreas, followed by 14 days of Usual Care. There was no washout period between arms.
  Bionic Pancreas: 14 days using the insulin-only configuration of the iLet Bionic Pancreas (Beta Bionics, Inc.), which automates insulin delivery, as the only intended mode of insulin delivery.
- PC Between Arms; EN Between Arms: Participants had up to 14 days from the stop of Arm 1 to schedule the start of Arm 2. This was not a washout period.
Arm/Group | PC Pre-randomization | EN Pre-randomization | PC-IP-UC | PC-IP-BP | PC-TH-UC | PC-TH-BP | EN-IP-UC | EN-IP-BP | EN-TH-UC | EN-TH-BP | PC Between Arms | EN Between Arms
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/9 | 0/10 | 0/10 | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 2/20 | 0/10 | 0/10 | 0/10 | 0/10 | 1/10 | 0/9 | 0/10 | 0/10 | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 5/20 | 2/20 | 0/10 | 2/10 | 1/10 | 2/10 | 2/10 | 0/9 | 3/10 | 0/10 | 0/20 | 1/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PC Pre-randomization (N=20) | EN Pre-randomization (N=20) | PC-IP-UC (N=10) | PC-IP-BP (N=10) | PC-TH-UC (N=10) | PC-TH-BP (N=10) | EN-IP-UC (N=10) | EN-IP-BP (N=9) | EN-TH-UC (N=10) | EN-TH-BP (N=10) | PC Between Arms (N=20) | EN Between Arms (N=19)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Not related to diabetes.
Severe hypoglycemia (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess in right axilla (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PC Pre-randomization (N=20) | EN Pre-randomization (N=20) | PC-IP-UC (N=10) | PC-IP-BP (N=10) | PC-TH-UC (N=10) | PC-TH-BP (N=10) | EN-IP-UC (N=10) | EN-IP-BP (N=9) | EN-TH-UC (N=10) | EN-TH-BP (N=10) | PC Between Arms (N=20) | EN Between Arms (N=19)
Hyperglycemia (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sinus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Acute phase reaction caused by Reclast
Illness/Cold/Flu (General disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carpal tunnel surgery (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatofibroma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract Surgery (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-27): https://cdn.clinicaltrials.gov/large-docs/57/NCT05168657/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-15): https://cdn.clinicaltrials.gov/large-docs/57/NCT05168657/ICF_001.pdf